CLINICAL TRIAL: NCT02352519
Title: A Randomized Comparison of Ultrasound Guided Bilateral Rectus Sheath Block and Local Anesthetic Infiltration for Postoperative Pain Control in Children With Acute Appendicitis
Brief Title: A Comparison of UGBRS Block and Local Infiltration
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Yang Liu, Pediatric Anesthesiologist, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H28183
Record Dates: First submitted 2014-07-24; First posted 2015-02-02 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UGBRSB (Experimental): Under sterile conditions,the posterior rectus sheath will be identified by ultrasound, and an insulated 22 gauge 50 mm needle inserted till the tip is seen to be directly between the rectus abdominis muscle and the posterior rectus sheath. Bupivacaine 0.25% (0.2 ml/kg with maximum 5 ml in each side) will be injected observing the spread on the ultrasound image.
  Interventions: Procedure: UGBRSB
- Local infiltration (Active Comparator): In those patients randomized to the LAI group, the surgeon will perform infiltration of 0.5 ml/kg of 0.25% bupivacaine (maximum, 10 ml) around the incision.
  Interventions: Procedure: Local Infiltration

INTERVENTIONS:
Procedure: UGBRSB — Under sterile conditions,the posterior rectus sheath will be identified by ultrasound, and an insulated 22 gauge 50 mm needle inserted till the tip is seen to be directly between the rectus abdominis muscle and the posterior rectus sheath. Bupivacaine 0.25% (0.2 ml/kg with maximum 5 ml in each side) will be injected observing the spread on the ultrasound image.
  Other Names: Ultrasound Guided Bilateral Rectus Sheath Block
  Arms: UGBRSB
Procedure: Local Infiltration — In those patients randomized to the LAI group, the surgeon will perform infiltration of 0.5 ml/kg of 0.25% bupivacaine (maximum, 10 ml) around the incision
  Other Names: Local Anesthetic Infiltration
  Arms: Local infiltration

SUMMARY:
In this research study, the investigators are trying to find out which of the two methods of injecting local anesthetics (at the site of the belly button cut or by ultrasound guided rectus sheath block) will provide better pain relief and less need for pain medication after surgery in children undergoing single incision laparoscopic appendectomy.

DETAILED DESCRIPTION:
Laparoscopic appendectomy is a common procedure in pediatric surgery. For single incision laparoscopic appendectomy (SILA), the laparoscope and other instruments are inserted with the aid of a large trocar through a single umbilical incision. Laparoscopic appendectomy via a single umbilical incision is a less invasive procedure associated with minimal or no scarring compared to the traditional laparoscopic operation. Postoperative pain, nausea and vomiting are common problems encountered with laparoscopic appendectomy and other abdominal operations. As an established standard practice at Texas Children's Hospital, pain control in these patients is achieved by intravenous opioids via a patient controlled device along with ketorolac tromethamine, as well as local anesthetic infiltration (LAI) performed by surgeon or bilateral rectus sheath blocks as described below.

The umbilical area is innervated by the bilateral 9th, 10th and 11th intercostal nerves, which run between the internal oblique and transversus abdominis muscle. At the lateral edge of the rectus muscle, the nerves perforate the rectus sheath and innervate the rectus muscle. Anterior cutaneous branches cross the muscle supplying the skin of the umbilical area. Successful blockade of the relevant intercostal nerves within the rectus sheath can provide effective pain relief for umbilical and other midline surgical incisions. Rectus sheath block has also been shown to give better pain control when compared with intra-incisional infiltration and intra-peritoneal injection in patients undergoing laparoscopic gynecologic surgery. Recently, it has been shown that there is improved efficacy and a decreased local anesthetic requirement when ultrasound is used to guide rectus sheath block in children undergoing umbilical hernia repair. However, data comparing pain after ultrasound guided bilateral rectus sheath block (UGBRSB) and peri-umbilical local anesthetic infiltration (LAI) for SILA are not available. The incidence of postoperative nausea and vomiting (PONV) is high after laparoscopic surgery, with a dose-related increase noted when opioids are used in the postoperative period. Effective regional anesthesia may decrease opioids use and consequently reduce the incidence of PONV and improve patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 1) Acute appendicitis (2) Age 6 - 17 years (3) American Society of Anesthesiologists Physical Status I - III (4) Patients undergoing SILA procedure performed by a single pediatric surgeon (Dr. Ashwin P. Pimpalwar) (5) Patients judged by parents, physicians and other caretakers as being capable of using the patient controlled analgesia (PCA) device.

Exclusion Criteria:

* 1) Patients who are not scheduled to undergo the procedure of SILA. (2) Patients with allergies to local anesthetics (3) Patients who do not understand or cannot use the pain rating scale because of developmental delay, language or other issues. (4) Patients with concomitant major cardio-respiratory disorders. (5) Patients judged to be incapable of using the PCA device (6) Patients who refuse to participate in the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Comparing the amount of morphine used during the first 48 hurs after surgery | 48 hours

SECONDARY OUTCOMES:
Comparing pain scores during the first 48 hours after surgery | 48 hours
Comparing time to first rescue analgesia | 48 hours
Comparing rescue analgesia used in the Post Anesthetic Care Unit (PACU) | 48 hours
Comparing incidence of side effects of opioids such as respiratory depression, itching, nausea, and vomiting, dysphoria | 48 hours
Comparing time to achieving discharge readiness in PACU | 48 hours
Comparing time to achieving discharge rediness from the hospital | 48 hours
comparing patient and parental satisfaction with pain management | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yang Liu, M.D>, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States